CLINICAL TRIAL: NCT02249351
Title: Efficacy and Safety of 48 mg Talsaclidine (Free Base) Tid po (Panel 1) and 60 mg Talsaclidine (Free Base) Tid po (Panel 2) for 12 Weeks in a Double-blind, Randomised, Placebo-controlled Within Escalating Dose Panels in 150 Patients With Mild to Moderate Dementia of Alzheimer Type
Brief Title: Efficacy and Safety of Talsaclidine (Free Base) in Patients With Mild to Moderate Dementia of Alzheimer Type
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506.209
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — talsaclidine fumarate

ARMS (2):
- Talsaclidine (Experimental)
  Interventions: Drug: Talsaclidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talsaclidine
  Arms: Talsaclidine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess symptomatic efficacy, safety and tolerability of talsaclidine in patients with mild to moderate dementia of Alzheimer type

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, age: over 40 years (lower age if genetic Dementia of Alzheimer Type (DAT) is documented). Patients over 85 years need to be in a clinically stable state (investigator's judgement)
* Patient's educational level is > 4 years
* Patient is able to understand the patient information and give informed consent
* Patient has given written informed consent in accordance with Good Clinical Practice and local legislation
* Patient has a relative or caregiver who is willing and capable to support the clinical trial; his/her written informed consent is optional
* Body weight: ≥ 50 kg and within +/- 30% of normal weight (Broca index)
* Diagnosis of DAT by the National Institute of Neurological and communicative Disorders-Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA) criteria
* MMS-score 10 - 24 inclusive
* Rosen ischemia score is lower or equal to two
* Patient is able to complete the trial examinations, to hear, speak, read and write in a basic way and primary sensorial functions are intact

Exclusion Criteria:

* Any dementia of vascular genesis (Rosen ischemia score > 2)
* Magnetic Resonance Imaging (MRI) or Computer Tomogram (CT) findings make the diagnosis of DAT unlikely (with a scan performed within 12 months of study entry)
* Any stroke history
* All secondary dementia (exclusion diagnosis defined by the NINCDS-ADRDA criteria) as a late complication of:

  * Cranio-cerebral trauma
  * Intoxication (incl. history of alcohol and drug abuse)
  * Cerebral infections (e.g. neurosyphilis)
  * Thyroid dysfunction
* Cerebral dysfunction due to metabolic disorders
* Possible reversible dementias secondary to a deficiency of vitamin B12, folic acid or thyroid hormone. Replacement therapy must be started three months before visit 1 in order to exclude dementia due to these deficiencies.
* Brain tumour (benign tumours found on CT not felt to be clinically relevant may be included, i.e.: meningioma)
* Down's syndrome, Parkinson's disease, Huntington's chorea, Diffuse Lewy Body Disease (as measured by the McKeith Criteria and specified in CTM)
* Multiple sclerosis
* Major depression with a score of <=16 on the Hamilton Depression Rating Scale (HAMD) 17 item scale
* Depressive pseudodementia
* Mental retardation
* Hydrocephalus
* Epilepsy
* Endogenous psychoses (schizophrenia)
* Untreated or poorly compensated hypertension (Blood Pressure systolic > 180 and/or diastolic > 110 mmHg)
* Hypertension being treated with reserpine, clonidine or β-blockers
* Severe heart disease (NYHA: III and IV)
* Any cardiac arrhythmias (atrial or ventricular) including bradycardia with a rate of < 50 bpm, arrhythmias due to second or third degree blocks and Lown: II-IV, Electrocardiogram > 30 ventricular extrasystoles/hour, multifocal or multiform and repetitive forms of ventricular extrasystoles, pacemakers are allowed
* Bronchial asthma with phases of exacerbation, or inducible by aspirin or other Nonsteroidal anti-inflammatory drugs, requiring acute pharmacologic intervention during the previous year
* Diabetes, type I or II, under active treatment with either insulin or an oral agent, diabetes controlled by diet and exercise alone is not excluded
* Renal insufficiency with a calculated creatinine clearance of less than 50 ml/min
* Abnormal urinalysis results as defined by:

  * a bacterial colony count of greater than 100,000/ml or
  * more than 10 leukocytes per high power field with more than 2 granular casts per low power field or
  * more than 10 red blood cells per high power field or
  * proteinuria >+ 1 (equivalent to > 30 mg/dl) and with a ratio of urine protein/urine creatinine > 0.3
* History of chronic urinary tract infection or recent urinary tract infection over the past six months
* History of renal stones within the past six months
* Acute hepatic disorder (liver enzymes above 50 % upper normal limit)
* Chronic hepatitis within the last two years (positive hepatitis titer, Hepatitis A Virus, Hepatitis B Virus, Hepatitis C Virus, cytomegalovirus, Epstein-Barr virus or abnormal immunological values (positive immunoglobulin M(IgM)/IgG) are allowed if all liver enzymes are within the normal range)
* History of liver disease within 2 years secondary to drug intoxication of any cause including drug intoxication (e.g. narcotics, cytostatics etc.)
* Patients with obvious symptoms of dehydration
* Abuse or dependence on drugs or other hepatotoxic agents by history or drug screen. A history of alcohol abuse within the last 10 years will also exclude the patient
* Neoplasm currently active or likely to recur, or in need of treatment (except basal cell carcinoma)
* Participation in another clinical trial within the last four weeks, or previous participation in a talsaclidine trial; patients who have been entered into panel 1 are not eligible for inclusion in panel 2
* Pregnant and lactating woman, woman with childbearing potential not using an approved method of contraception
* Poor ability of the patient or caregiver/family to comply with protocol requirements as assessed by the investigator
* A list of excluded medications is attached to the protocol. These medications have to be replaced at least four weeks before the trial medication is started. If replacement in not clinically advisable, then the patient has to be excluded from the trial
* In Germany, patients with the following additional diagnosis are excluded

  * manifest angina pectoris as well as
  * peripheral arterial circulatory disturbances

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1999-12; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive part (ADAScog) | Baseline, week 4, 8, 12

SECONDARY OUTCOMES:
Change in ADAScog (extension) | Baseline, week 4, 8, 12
Change in ADAScog (Total) | Baseline, week 4, 8, 12
  Defined as ADAScog + ADAScog(extension)
Change in mini mental state (MMS) | Screening, week 12
Change in neuropsychiatric inventory (NP) | Baseline, week 12
Change in Hamilton Depression Rating Scale (HAMD 17 item scale) | Screening, week 12
Change in instrumental activity of daily living (IADL) | Baseline, week 12
Change in living status rated on a 6-point scale | Baseline, week 12
Change in clinician's global impression rated with Alzheimer's Disease cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | Baseline, week 12
Number of patients with adverse events | up to 6 months